CLINICAL TRIAL: NCT04107038
Title: A Randomized Controlled Trial Comparing Monitored Anesthesia Care Versus General Anesthesia With Transesophgeal Echocardiography for Transcatheter Aortic Valve Replacement
Brief Title: Monitored Anesthesia Care vs. General Anesthesia for Transcatheter Aortic Valve Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, George Whitener, Principal Investigator, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00088473
Record Dates: First submitted 2019-09-11; First posted 2019-09-27 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Transcatheter Aortic Valve Replacement
Keywords: Anesthesia, TAVR, Cardiothoracic, Cardiology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- General (Active Comparator): Participants randomized to group A will receive general endotracheal anesthesia as their anesthetic procedure.
  Interventions: Procedure: General Endotracheal Anesthesia
- Sedation (Active Comparator): Participants randomized to group B will receive monitored anesthesia care as their anesthetic procedure.
  Interventions: Procedure: Monitored anesthesia care

INTERVENTIONS:
Procedure: General Endotracheal Anesthesia — Participants receive general endotracheal anesthesia for the procedure, as well as analyzing the information from their transesophageal echocardiography per routine clinical care.
  Arms: General
Procedure: Monitored anesthesia care — Participants receive monitored anesthesia care for their procedure.
  Arms: Sedation

SUMMARY:
This study is being done to evaluate the impact that monitored anesthetic care (MAC) versus general endotracheal anesthesia (GETA) has on hospital length of stay, rate of ICU admission, and procedural mortality for patients undergoing Transcatheter Aortic Valve Replacement (TAVR). Also, the investigators hope to determine if the use of Transesophageal Echocardiography (TEE) during GETA impacts device success. Adult patients undergoing transfemoral approach TAVR for aortic valve stenosis may be eligible candidates for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥ 18 years old
* Adult patients undergoing transfemoral approach TAVR for aortic valve stenosis
* Adult patients who are medically eligible to receive both anesthetics (GA and MAC)

Exclusion Criteria:

* Inability to speak English
* Body Mass Index (BMI) > 37 kg/m2
* History of difficult airway requiring fiberoptic intubation
* Inability to lie flat
* Women who are pregnant
* Patients who have contraindications to either anesthetic, such as an allergy or history of malignant hyperthermia, will also be excluded from the study.
* Inability or unwillingness of subject to give informed consent based on any reason
* Patients with any of the following absolute contraindications to TEE:
* Perforated Viscus
* Esophageal Stricture
* Esophageal Tumor
* Esophageal Perforation
* Esophageal Diverticulum
* Active upper GI Bleed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Hospital Length of Stay | Up to 1 month
  The total number of hours that the patient stayed in the hospital will be measured from the "Anesthesia Start" time until their time of discharge, as recorded in their electronic medical record.
ICU Admission Rate | Up to 48 hours
  The investigators will determine the ICU admission rate by taking the total number of patients admitted to the ICU and dividing it by the number of cases in each arm of the study, based on MUSC's "fast track" pathway and our inclusion.
Procedural Mortality | Up to 30 days
  The percentage of the study population that died within 30 days of their procedure or during index procedure hospitalization - if the postoperative length of stay is longer than 30 days.

SECONDARY OUTCOMES:
Paravalvular Regurgitation | For GETA cases, will be recorded after valve implantation. For all cases, will be recorded from a TTE report that is completed on post-operative day 1 or 2 and at 1 year.
  Paravalvular regurgitation is a specific type of aortic regurgitation that is determined qualitatively by the echocardiographer. It is defined as the grade of aortic valve regurgitation around the perimeter of the implanted prosthesis. The assigned grade will be classified according to a unifying five-class scheme, at the determination of the cardiologist. Grade of aortic regurgitation is measured as none, mild, moderate, or severe. None is best, severe is worst. For GETA cases, paravalvular regurgitation will be recorded after valve implantation by the anesthesiologist performing TEE, as is routine. For all cases, paravalvular regurgitation will be recorded from a TTE report that is completed on post-operative day 1 or 2 (the 1st post-operative TTE) during routine clinical care, and again by TTE report at 1 year during routine clinical follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: George Whitener, M.D., Principal Investigator — Medical University of South Carolina - Department of Anesthesia
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No